CLINICAL TRIAL: NCT03657225
Title: Comparison Of Mini-Bypass To Conventional Cardiopulmonary Bypass In Asian Patients Undergoing Coronary Artery Bypass Grafting Surgery
Brief Title: Mini Versus Conventional Cardiopulmonary Bypass In CABG in Asian Patients
Acronym: MiniCPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHG DSRB 2008/00332
Record Dates: First submitted 2014-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Acute Kidney Injury; Neurological Injury
Keywords: miniaturized; cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury; Trauma, Nervous System

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini CPB (ECCO, Sorin, Italy) (Active Comparator): Utilization of the mini CPB circuit (Extra Corporeal Circuit Optimized; Phisio, Sorin Group, Italy)
  Interventions: Device: Utilization of the mini CPB circuit
- Conventional (Placebo Comparator): Use of conventional CPB circuit
  Interventions: Drug: Utilization of the conventional circuit

INTERVENTIONS:
Device: Utilization of the mini CPB circuit — Comparison of the mini CPB circuit to conventional circuit
  Arms: Mini CPB (ECCO, Sorin, Italy)
Drug: Utilization of the conventional circuit — Comparison of the mini CPB circuit to conventional circuit
  Arms: Conventional

SUMMARY:
Our intention is to perform a randomized controlled trial to compare the efficacy and safety of mini cardiopulmonary bypass system to a modified conventional bypass circuit in 80 Asian patients undergoing elective CABG. Our intend is to confirm the efficacy of mini-bypass in reducing haemodilution and reducing blood transfusions, and investigate if this is associated with reduced inflammation and better cardiovascular, neurological, renal, respiratory and infection outcome.

DETAILED DESCRIPTION:
Mini-bypass systems have the potential to reduce the problems associated with conventional cardiopulmonary bypass systems by preserving hematocrit, reducing transfusion requirements, and reducing inflammation. Intuitively, this system would be ideal for our smaller Asian patients, who as a result of their body sizes, are prone to severe hemodilution and increased transfusion requirements. However, our initial results based on established Western protocols were not as good as the investigators hoped. Using a modified protocol, the investigators were able to reduce perioperative blood transfusion. Therefore, the investigators intend to prospectively confirm the efficacy of mini-bypass in conjunction with our modified protocol in reducing haemodilution and reducing blood transfusions. The investigators will also establish the safety of this protocol, and investigate if this is associated with reduced inflammation and better cardiovascular, neurological, renal, respiratory and infection outcomes.

80 Asian patients undergoing primary coronary artery bypass grafting with cardiopulmonary bypass will be randomly divided either to utilize the mini-bypass system (Extra Corporeal Circuit Optimized; Phisio, Sorin Group, Italy) or the conventional system. Anaesthesia, surgical and perfusion management will be standardized, except for measures specific to the establishment of mini-bypass. The primary outcome measures will be haemodilution (first and lowest hematocrit) during cardiopulmonary bypass, blood loss in the first 24 and 48 hours post-operatively, and perioperative blood transfusions. Secondary outcomes include safety profile (air embolization, hypoperfusion), inflammation (TNF-alpha, interleukin-6, C-reactive protein, lactate dehydrogenase) in the first 72 hours after bypass, clinical outcomes (renal, neurological, cardiac, respiratory) and resource utilization (blood utilization, length of stay).

This project will allow us to confirm our retrospective findings that mini-bypass systems in conjunction with our modified protocol will benefit our smaller patients haematologically and lead to tremendous savings in blood utilization. The investigators will also establish if this protocol is safe, and if there are additional benefits in terms of inflammation, clinical outcomes and resource utilization. Our findings will also be applicable throughout East Asia, as patients in the region generally lag our Western counterparts in size.

ELIGIBILITY:
Inclusion Criteria:

* first time on pump CABG revascularization

Exclusion Criteria:

* poor left ventricular ejection faction (< 30%)
* immunologic disease or malignancies
* acute inﬂammatory disease
* coagulopathy
* steroid treatment
* preoperative renal failure (currently receiving dialysis)
* significant carotid disease

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 48 hours after surgery
  Meeting AKIN 1 criteria

SECONDARY OUTCOMES:
Neurocognitive decline | 3 months post surgery
  Use of Neurocognitive test / questionnaire: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Inflammation | 72 hours post surgery
  Markers for inflammation will be measured preoperatively, and daily till the 3rd postoperative day, including TNF-alpha, IL-6 and C-Reactive Protein.

OTHER OUTCOMES:
Atrial fibrillation | 7 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lian K Ti, MBBS, MMed, Principal Investigator — National University Health System, Singapore
Locations (1):
- National University Health System, Singapore, Singapore

REFERENCES:
- [Background] Ti LK, Goh BL, Wong PS, Ong P, Goh SG, Lee CN. Comparison of mini-cardiopulmonary bypass system with air-purge device to conventional bypass system. Ann Thorac Surg. 2008 Mar;85(3):994-1000. doi: 10.1016/j.athoracsur.2007.09.001. PMID 18291186